CLINICAL TRIAL: NCT04592848
Title: Female Sexual Function and Sexual Quality of Life After Cystectomy or Urinary Diversion in Patients With Non-malignant Disease
Brief Title: Female Sexual Function After Cystectomy
Acronym: FSFAC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0873
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Sexual Activity
MeSH Terms: conditions — Sexual Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population study: Female patients who undergone a cystectomy and/or urinary diversion for a non-malignant disease at "Lyon Sud" Hospital between January 2007 and December 2019.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Four Questionnaires in French will be sent to participants :
  * 1 questionnaire about sexual and urinary symptoms before and after the surgery ;
  * 1 validated questionnaire "Female Sexual Function Index" to assess sexual function over the past 4 weeks ;
  * 1 validated questionnaire "Body Image Scale" to assess body image during the past week ;
  * 1 validated questionnaire "Stoma Quality of Life", only for patients with incontinent urostomy.
  If the questionnaires are not returned 15 days after sending, a follow-up phone call will be made by one of the investigators.
  The data collection will include both the answers to the questionnaires and the patients' computerized medical data:
  * Pathology responsible for the urological disorders and date of onset of the disorders
  * Date and Type of surgery performed
  * Patient's age at the time of surgery
  * Post-operative complications within one month of surgery

SUMMARY:
Cystectomy with bladder replacement, with or without urinary diversion, is the preferred treatment option for benign pathologies responsible for neurogenic bladder or sphincter dysfunction after failure of conservative treatments.

This surgery has both the objective of preventing urological complications and improving quality of life.

We know that women are especially affected by these conditions, as demonstrated by the high prevalence of demyelinating diseases such as multiple sclerosis in this population. Patients are often young and sexually active before the surgery.

Despite the existence of validated evaluation tools since the early nineties, there is poor data exploring effects of invasive procedures such as cystectomy on sexual activity and quality of sexual life in female patients.

Indeed, existing literature largely focuses on sexual function in male population after cystectomy for urothelial cancer.

Data on sexual function after stoma formation in women with colorectal cancer show a significant change after the surgery, partly due to body image issues. We can easily suppose that there's also an important impact of cystectomy that may affect sexual quality of life.

Thus, the objective of the study is to assess sexual function and determine factors that may influence sexual quality of life in female patients following cystectomy or urinary diversion.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged from 18 to 75 years
* With Partial or total cystectomy and/or urinary diversion and/or urinary ostomy repair operations between 01/01/2007 and 15/12/2019 at the "Lyon Sud" Hospital.
* Surgery was performed for urological disorders caused by a non-malignant disease
* Patients currently more than 6 months away from the last urological cystectomy/ urinary diversion/ urinary stoma repair surgery

Exclusion Criteria:

* Patients deceased
* Patients who undergone a partial cystectomy without urinary diversion for endometriosis with bladder involvement
* Patients unable to complete the questionnaires

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists in alive female patients aged 18-75 years, who undergone a partial or total cystectomy and/or urinary diversion and/or urinary ostomy repair operations between 01/01/2007 and 15/12/2019 at the "Lyon Sud" Hospital and able to complete the questionnaires.
  All patients suffer from urological disorders caused by a non-malignant pathology, and have had surgery after failure of conservative therapies.
  Among the patients identified from the computerized medical records, 55 suffer from Multiple sclerosis, 29 patients from Spinal Cord Injury, 21 suffer from Suprapontine and pontine lesion or disease, 19 suffer from non-traumatic lesion or disease between caudal brainstem and sacral spinal cord,18 suffer from lesions of the peripheral nervous system, 8 suffer from interstitial cystitis or idiopathic disorders and 1 suffers from a neurodegenerative disease of unknown etiology
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
FSFI Total Score in study population | at least 6 months after the surgery (Cystectomy and/or urinary diversion)
  The FSFI Score will be obtained from answers of the validated questionnaire "Female Sexual Function Index", a 19-item self-report measure of female sexual function.
  It uses a 5-point Likert scale ranging from 1-5 for each item. It provides scores on overall levels of sexual function and its six components: Desire, Arousal, Lubrication, Orgasm, Satisfaction and Pain. The full scale score is between 2 and 36.
  According to literature, total score of 26 or less indicates a risk of sexual dysfunction.
  The version used in this study is the French one.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud (Hospices Civils de Lyon), Pierre-Bénite, France